CLINICAL TRIAL: NCT07347483
Title: Assessment of Trunk Position Sense, Trunk Control, and Functional Independence in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Selvin BALKİ, Assoc. prof. Dr, Cumhuriyet University
Other Study IDs: SCU-FTR-SB-04
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
Keywords: Trunk Position Sense; Trunk Control; Functional Independence; Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spastic Cerebral Palsy
  Interventions: Other: Only measurements were taken.

INTERVENTIONS:
Other: Only measurements were taken. — This study does not contain any intervention.

SUMMARY:
The purpose of this study is to determine whether there is a difference in trunk proprioception, as assessed by trunk position sense, in children with unilateral and bilateral spastic cerebral palsy, and to evaluate the relationship between trunk position sense, trunk control, and functional independence.

DETAILED DESCRIPTION:
This cross-sectional and descriptive study was conducted in children with unilateral and bilateral spastic cerebral palsy aged between 6 and 12 years. A total of 78 children (36 girls and 42 boys) with spastic cerebral palsy were included in the study. The gross motor function levels of the participants ranged from Level I to Level IV according to the Gross Motor Function Classification System (GMFCS).

Participants were recruited from children receiving education and rehabilitation services at special education and rehabilitation centers in Kayseri, Turkiye, and only children whose parents or legal guardians provided written informed consent were included.

Demographic and clinical characteristics of the participants were recorded using a structured sociodemographic data form.

Trunk position sense was assessed using a dual inclinometer device to evaluate trunk proprioception. Trunk control was evaluated using the Trunk Impairment Scale, and functional independence was assessed using the motor subscale of the Pediatric Functional Independence Measure (WeeFIM). In addition, muscle tone was assessed bilaterally using the Modified Ashworth Scale.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of unilateral or bilateral spastic cerebral palsy,
* Are aged between 6 and 12 years,
* Are able to sit independently,
* Have a cognitive level sufficient to understand and follow verbal instructions,
* Have not undergone surgical intervention or Botulinum Toxin A injection within the last 6 months,
* Have parents or legal guardians who have provided written informed consent.

Exclusion Criteria:

* Have received Botulinum Toxin or intrathecal baclofen treatment within the last 6 months,
* Have a history of pelvic, spinal, or upper extremity surgery,
* Have severe visual or hearing impairments,
* Have cognitive impairments preventing effective communication,
* Are unable to sit independently,
* Do not have parental consent.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Spastic cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Trunk Position Sense | Data collection was conducted between January 2022 and March 2023.
  Trunk proprioception assessed using a dual inclinometer device during trunk flexion movements with the repositioning angle method under eyes-open and eyes-closed conditions.

SECONDARY OUTCOMES:
Trunk Control | January 2022 - March 2023
  Assessed using the Trunk Impairment Scale (TIS) in sitting position.
Functional Independence | January 2022 - March 2023
  Assessed using the motor subscale of the Pediatric Functional Independence Measure (WeeFIM).
Muscle Tone | January 2022 - March 2023
  Assessed bilaterally using the Modified Ashworth Scale (MAS).

CONTACTS AND LOCATIONS:
Overall Officials: Selvin Balki, Assoc. prof. Dr, Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No